CLINICAL TRIAL: NCT05979194
Title: WHO Labour Care Guide Introduction, Implementation and Use as an Effective Decision-making Tool to Monitor Labor Among Obstetric Care Providers in Publicly Funded Health Facilities in Mbarara District and Mbarara City, Southwestern Uganda
Brief Title: WHO Labor Care Guide for Obstetric Care Providers in Public Health Facilities in Mbarara, Southwestern Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REC2023
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Intrapartum Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Labor care guide (Other): In this study, we shall determine the effectiveness and other implementation outcomes of the new LCG using Proctor implementation outcome framework among HCPs delivering women across Mbarara District and Mbarara City and evaluate the diagnostic accuracy of the new WHO LCG versus the partogram in detecting prolonged labour and reducing rates of obstructed labour among women delivering in Mbarara district. We shall use local contextualized data from qualitative one-on-one key informant interviews in objective 1 from HCPs and Ministry of Health official involved in labour monitoring and implementation. The WHO labour care guide shall be refined and a Ugandan Ministry of Health prototype designed. An appropriated training and implementation strategy informed by the HCPs themselves shall be used to deliver the content to HCPs in all pilot sites.
  Interventions: Behavioral: Labor Care Guide

INTERVENTIONS:
Behavioral: Labor Care Guide — Identifying information and labor characteristics at admission, supportive care, care of the baby, care of the woman, labor progress, medication, and shared decision-making

SUMMARY:
The goal of this mixed method multisite effectiveness-implementation study across all basic and comprehensive emergency obstetric and newborn care facilities in Mbarara district and Mbarara City in Southwestern Uganda is to identify unique challenges, facilitators and patterns of potential and sustained uptake of the new WHO Labor Care Guide. Using these baseline findings, I will characterize, and refine the LCG, and then develop a suitable training strategy to effectively integrate/implement the new LCG into routine maternity care in Mbarara district. I will then utilize the Proctor implementation outcome framework to evaluate implementation outcomes of using the new labor care guide in routine maternity care that include; acceptability, appropriateness, feasibility, fidelity, and effectiveness among HCPs actively involved in deliveries across Mbarara District and Mbarara City. Finally, I will assess the diagnostic predictability of the new LCG compared to the partogram in effectively detecting prolonged labor among women delivering in Mbarara district and Mbarara City.

DETAILED DESCRIPTION:
I will utilize an ambispective cohort; a combination of a historical cohort of mothers monitored using a partograph and prospective cohort of women monitored using the new Labor Care Guide to evaluate implementation success (effectiveness). As a concerted effort to meaningfully implement a new intervention meant to reduce preventable maternal and perinatal morbidity and mortality, these results will generate grounded, robust scientific data to inform stakeholders and policy makers working towards effectively integrating and scaling up of this new LCG into routine maternity care in similar settings across the country and beyond. This study will also be able to show the effect of this intervention, and optimize its implementation in routine maternity care practice to improve maternal-fetal outcomes in similar settings.

Participants will be adult HCPs actively involved in maternity care and conducting deliveries, health facility managers in Mbarara district and officials from the reproductive health division of the Ugandan Ministry of Health. For the effectiveness-implementation trial, we shall enroll 520 mothers in active labor at the study facilities. Abstracted partograph data from the records of 520 mothers whose labor was monitored using partograph data will be used to compare the proportion of prolonged labor in addition to other effectiveness outcomes.

The main questions we aim

* To determine the effectiveness and other implementation outcomes of the new LCG using Proctor implementation outcome framework among HCPs delivering women across Mbarara District and Mbarara City and
* To evaluate the diagnostic accuracy of the new WHO LCG versus the partogram in detecting prolonged labor and reducing rates of obstructed labor among women delivering in Mbarara district Adult HCPs will participate in audio recorded in-dept face to face interviews and adult mothers in labor will be monitored using the New WHO labor care guide to document the proportion of prolonged labor defined as 1) labor crossing the action line on the partograph and 2) labor lasting more than a specified centimeter cervical dilation "time lag" in the alert column of section 5 of the LCG. Secondary outcome measurements will include proportion of obstetric interventions such as caesarean sections, labor augmentation, blood transfusion; quality-of-care; having a fresh still birth; duration of 1st and 2ndstages of labor; 5-minute apgar score, need for resuscitation /blood transfusion, mode of delivery; initiation of breastfeeding; obstetric complications diagnosed and or managed during labor, childbirth or immediate postpartum; ruptured uterus; postpartum hemorrhage; maternal/newborn sepsis; maternal, fetal, and newborn deaths. Other quantitative data that will be collected from maternity records of women that have delivered within one year before and a year after implementation of the labor care guide will include; patient demographics e.g., age, gravidity, parity, gestational age, prenatal, antepartum high-risk morbidities, NCDs, and HCP demographics; age, education, experience, self-efficacy will be collected

ELIGIBILITY:
Inclusion Criteria:

* Individuals with self-reported willingness to use the new LCG in monitoring of labor, able and willing to provide informed consent will be invited to participate in this study.

Exclusion Criteria:

* Individuals unwilling to use the LCG and unable to provide informed consent will not be eligible to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with prolonged labor | 6 months
  We will define prolonged labor as 1) labor crossing the action line on the partograph, 2) labor lasting more than a specified centimeter cervical dilation "time lag" in the alert column of section 5 of the LCG

SECONDARY OUTCOMES:
Proportion of obstetric interventions | 6months
  proportion of obstetric interventions such as caesarean sections, labour augmentation, blood transfusion; quality-of-care; having a fresh still birth; duration of 1st and 2nd stages of labor; 5-minute apgar score, need for rescuscitation/blood transfusion, mode of delivery; initiation of breastfeeding; obstetric complications diagnosed and or managed during labor, childbirth or immediate postpartum; ruptured uterus; postpartum hemorrhage; maternal/newborn sepsis; maternal, fetal, and newborn deaths

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Mugyenyi, MMed, Principal Investigator — Mbarara University of Science and Technology

REFERENCES:
- [Derived] Mugyenyi GR, Tumuhimbise W, Atukunda EC, Tibaijuka L, Ngonzi J, Kayondo M, Kanyesigye M, Musimenta A, Yarine FT, Byamugisha JK. Effectiveness of the Modified WHO Labour Care Guide to Detect Prolonged and Obstructed Labour Among Women Admitted at Eight Publicly Funded, Midwife-Led Community Health Facilities in Rural Mbarara District, Southwestern Uganda: An Ambispective Cohort Study. Int J Womens Health. 2025 Feb 4;17:271-285. doi: 10.2147/IJWH.S498903. eCollection 2025. PMID 39925783
- [Derived] Godfrey MR, Wilson T, Esther AC, Leevan T, Joseph N, Musa K, Micheal K, Angella M, Fajardo YT, Josaphat BK. Effectiveness of the modified WHO labour care guide to detect prolonged and obstructed labour among women admitted at publicly funded facilities in rural Mbarara district, Southwestern Uganda: an ambispective cohort study. medRxiv [Preprint]. 2024 Sep 5:2024.09.04.24313073. doi: 10.1101/2024.09.04.24313073. PMID 39281732
- [Derived] Mugyenyi GR, Byamugisha J, Tumuhimbise W, Atukunda E, Yarine FT. Labour Care Guide implementation as a decision-making tool for monitoring labour among healthcare providers in Uganda: protocol for a mixed-methods study. BMJ Open. 2024 Apr 15;14(4):e079216. doi: 10.1136/bmjopen-2023-079216. PMID 38626961